CLINICAL TRIAL: NCT03586674
Title: Fibrates: An Adjuvant Therapy for Cholestasis In Pediatric Age Group
Brief Title: Fibrates in Pediatric Cholestasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoda A. Atta (Other Government)
Responsible Party: Sponsor-Investigator, Hoda A. Atta, Pediatric Specialist, Ministry of Health and Population, Egypt
Organization: Ministry of Health and Population, Egypt (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1984
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Chronic Cholestasis
Keywords: pediatric cholestasis, Fibrate
MeSH Terms: interventions — Fenofibrate; Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ursogal (Active Comparator): Control group : Ursogal 10-20 mg/kg/d on 2 divided dose for four months with regular follow up.
  Interventions: Drug: Ursogal
- Lipanthyl + Ursogal (Experimental): Therapy group: Ursogal 10-20 mg/kg/d by mouth, on 2 divided dose, and lipanthyl 10-20 mg/kg/d by mouth,once per day, for four months with regular follow up.
  Interventions: Drug: Lipanthyl; Drug: Ursogal

INTERVENTIONS:
Drug: Lipanthyl — Tablet
  Other Names: ursogal
  Arms: Lipanthyl + Ursogal
Drug: Ursogal — suspension
  Other Names: non

SUMMARY:
A study conducted to assess the effect of fibrates on pruritus and biochemical picture in pediatric patients with cholestatic liver diseases.

DETAILED DESCRIPTION:
Cholestatic liver disorders include a spectrum of hepatobiliary diseases of diverse etiologies that are characterized by impaired hepatocellular secretion of bile, resulting in accumulation of bile acids, bilirubin and cholesterol.This could result in different clinical features including pruritus, malabsorption and vitamin deficiencies with subsequent coagulation disorders and bone disease. Persistence of cholestasis leads to biliary fibrosis which can progress to liver cirrhosis and end-stage liver disease.

Nuclear receptors (NRs) regulate ligand-activated transcription factor networks of genes for the elimination and detoxification of potentially toxic biliary constituents accumulating in cholestasis. Activation of several NRs also modulates fibrogenesis, inflammation, and carcinogenesis as sequelae of cholestasis. Hence, It represent attractive targets for pharmacotherapy of cholestatic disorders.

Several already available drugs may exert their beneficial effects in cholestasis via NR activation eg, ursodeoxycholic acid via glucocorticoid receptor and pregnane X receptor, and rifampicin via pregnane X receptor. Unfortunately, Some patients may not respond to these medications.

Fibrates, serum Lipid lowering medication, has a stimulation action on proliferator activated receptor alpha. It is a nuclear receptor with an integral role in bile homeostasis. Several case reports and pilot studies have demonstrated the efficacy of fibrates in reducing serum biomarkers of cholestasis and liver function abnormalities in patients with incomplete response to ursodeoxycholic acid monotherapy. These results are of interest, because fibrates are attracting increased attention as adjunct therapy for chronic cholestatic liver diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic cholestatic liver disease defined as any condition in which substances normally excreted into bile are retained for more than 6 months.

Exclusion Criteria:

* Patients with anatomical or mechanical obstructive causes for cholestasis.
* Cholestatic patients who were suffering from another liver disease.
* Cholestatic patients who were receiving drugs affecting lipid profile.
* Patients receiving drugs that interact with Fenofibrate (FF) e.g statins and warfarin
* Patients with non obstructive gall bladder stones were excluded from T gp.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Change in the pruritus grading score | four months
  The pruritus grading score includes four areas each has its score: distribution score 1-3;1= single site and 3 generalized, Severity score 1-5 ; 1= rubbing,5 = general excoriation, Frequency score 1-5; 1= episodic,5= continuous, and Sleep disturbance score 0-6 ; 0= no effect on sleep, 6= total restless.

SECONDARY OUTCOMES:
Changes in the liver function test and lipid profile | four months
  investigate the effect on Alanine Aminotransferase (ALT),Aspartate Aminotransferase (AST) ,Albumin,Bilirubin, Bile acid, lipid profile

CONTACTS AND LOCATIONS:
Overall Officials: Tawhida Y Abdel Ghaffar, MD, Study Director — ASU
Locations (2):
- Egypt (2):
  - Dr. Yassin Abdel Ghaffar Charity Center For Liver Diseases & Researches, Cairo, Nasr City
  - National liver istitute, Shibīn al Kawm

IPD SHARING:
Plan to Share IPD: No
Only overall results will be shared.

REFERENCES:
- [Background] Ghonem NS, Boyer JL. Fibrates as adjuvant therapy for chronic cholestatic liver disease: its time has come. Hepatology. 2013 May;57(5):1691-3. doi: 10.1002/hep.26155. Epub 2013 Apr 5. No abstract available. PMID 23174993
- See also: Review article — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4048949/